CLINICAL TRIAL: NCT05374226
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Recombinant Fully Human Anti-CD39 Monoclonal Antibody JS019 in Patients With Advanced Solid Tumors or Lymphomas
Brief Title: A Phase 1 Study to Evaluate JS019 in Advanced Solid Tumors or Lymphomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suzhou Kebo Ruijun Biotechnology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS019-001-I
Record Dates: First submitted 2022-05-05; First posted 2022-05-16 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-04

CONDITIONS: Advanced Solid Tumors or Lymphomas
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- JS019 0.3 mg/kg (Experimental): repeat dose every 21 days up
  Interventions: Biological: JS019
- JS019 1 mg/kg (Experimental): repeat dose every 21 days up
  Interventions: Biological: JS019
- JS019 3 mg/kg (Experimental): repeat dose every 21 days up
  Interventions: Biological: JS019
- JS019 10 mg/kg (Experimental): repeat dose every 21 days up
  Interventions: Biological: JS019

INTERVENTIONS:
Biological: JS019 — Four dose levels are preset: 0.3 mg/kg, 1 mg/kg, 3 mg/kg, and 10 mg/kg. The subjects are treated with JS019 by intravenous infusion, once every 3 weeks (Q3W). A treatment cycle is 21 days, and the DLT observation period is 21 days after the first administration.

SUMMARY:
This is a phase 1 clinical study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of JS019 as monotherapy in patients with advanced malignant solid tumors/lymphomas.

The study includes JS019 monotherapy dose escalation, dose expansion and indication expansion stages to investigate the safety, tolerability, pharmacokinetics and preliminary anti-tumor efficacy of JS019 as monotherapy.

DETAILED DESCRIPTION:
Monotherapy Dose Escalation Stage:

In this stage, the safety and tolerability, PK characteristics, immunogenicity and PD of JS019 are investigated. Four dose levels are preset: 0.3 mg/kg, 1 mg/kg, 3 mg/kg, and 10 mg/kg. The subjects are treated with JS019 by intravenous infusion, once every 3 weeks (Q3W). A treatment cycle is 21 days, and the DLT observation period is 21 days after the first administration. During the study, necessary adjustments may be made to the escalating dose and dosing interval based on the safety, PK and other results obtained.

Monotherapy Dose Expansion Stage:

SMC will select 1~2 dose levels (dose levels in the monotherapy dose escalation stage or intermediate dose levels) of JS019 as monotherapy. Each dose level includes 6~9 subjects with advanced malignancies to further evaluate the safety, pharmacokinetics, immunogenicity, pharmacodynamics and efficacy of JS019 as monotherapy, and determine the RP2D of JS019 as monotherapy.

Monotherapy Indication Expansion Stage Based on the determined RP2D of JS019 as monotherapy, 2-4 specific malignancies are selected for indication expansion; about 20-30 patients are included for each indication. It is planned to include expansion cohorts to explore the efficacy and safety of JS019 as monotherapy. The actual cohorts included may be adjusted based on the results of the previous studies.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and willing to sign the Informed Consent Form;
2. Male or female aged 18~75 years (included);
3. Patients with pathologically confirmed advanced malignant solid tumors or lymphomas;
4. Failed or unsuitable for standard treatment, received at least one line of systemic treatment;
5. Eastern Cooperative Oncology Group (ECOG) physical fitness score: 0~1;
6. Expected survival period ≥ 12 weeks;
7. At least one measurable lesion according to criteria RECIST v1.1 or Lugano 2014;

Exclusion Criteria:

1. Patients with known hypersensitivity to the components of JS019;
2. Patients who have received the treatment with anti-CD39 antibodies or inhibitors;
3. Patients who participated in other clinical studies within 4 weeks prior to the first administration of JS019, except patients are in the follow-up period of observational (non-interventional) clinical study or interventional study;
4. Patients who have received major surgery within 4 weeks before the first dose or expected to undergo major surgery during the study (as judged by the investigator) or are in the recovery period from surgery;
5. Patients who have received anti-tumor therapy, such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, or biological therapy, within 4 weeks or 5 half-lives of the therapy (whichever is shorter) prior to the first dose of JS019. Patients who have received traditional Chinese medicine or Chinese patent medicine preparations with anti-tumor indications within 2 weeks before the first dose of JS019. Can accept hormone therapy for non-tumor-related diseases (such as insulin therapy for diabetes and hormone replacement therapy, etc.);
6. Patients who have discontinued immunotherapy due to immune-related AEs.
7. Patients who have used immunosuppressive drugs within 4 weeks prior to the first dose of JS019, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids ≤10 mg/day prednisone or equivalent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2023-12-11 (Estimated); Study Completion 2024-03-07 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | 2 years
  Incidence of DLT, incidence and severity of adverse events (AEs) and serious adverse events (SAEs), clinically significant abnormal changes in laboratory tests and other tests
Maximum tolerated dose (MTD, if possible) and the recommended phase 2 dose (RP2D) | 2 years
  Maximum tolerated dose (MTD) : The highest dose at which <1/3 patients experience DLT events.
  Phase II recommended dose: safety, pharmacokinetics, and preliminary efficacy data of dose escalation will be integrated. When the Maximum tolerated dose(MTD) is determined, the Maximum tolerated dose(MTD) is usually used as the Phase II recommended dose(RP2D), or the dose lower than the Maximum tolerated dose(MTD) is selected as the Phase II recommended dose(RP2D) based on the comprehensive data.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | 2 years
  Drug concentrations in individual subjects at different time points after administration
Immunogenicity | 2 years
  Incidence of anti-drug antibodies (ADA), titer of ADA-positive samples.
Pharmacodynamics （PD） | 2 years
  CD39 receptor occupancy in peripheral blood.
Objective response rate (ORR) | 2 years
  The percentage of cases with remission (PR + CR) after treatment was assessable
Duration of response (DOR) | 2 years
  The time from the first assessment of CR or PR to the first assessment of PD or death due to any cause.
Disease control rate (DCR) | 2 years
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
Time to response (TTR) | 2 years
  time from the start of treatment to progression of diease.
Progression-free survival (PFS) | 2 years
  PFS is defined as time from the start of treatment to progression of disease or death.
Overall survival (OS) | 2 years
  Overall survival is defined as time from the start of treatment until death due to any reason.

OTHER OUTCOMES:
Biomarkers | 2 years
  The expression levels of CD39, P2X7, PD-L1 and CD8+ in tumor tissue, and the correlation between their expression levels and efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China